CLINICAL TRIAL: NCT05919901
Title: Multi-level School-based Intervention to Improve HPV Vaccine Uptake and Completion in South Africa
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The study is currently halted due to ongoing amendments following major protocol changes
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ingrid Theresa Katz, M.D., Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023p001246
Record Dates: First submitted 2023-06-12; First posted 2023-06-26 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: HPV

STUDY DESIGN:
Intervention Model Description: We will select 10 schools (~60 parents/children per school) by a stratified random sampling approach. We will randomize schools in a 1:1 ratio to the intervention and control arms. Randomization, based on a computer-generated assignment, will occur after the 10 schools have been selected. Control participants will be eligible to receive the intervention materials at the end of the 1-year follow-up period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HPV Intervention (Experimental)
  Interventions: Other: HPV Vaccine Communication Strategy
- Active Control (Active Comparator)
  Interventions: Other: HPV Vaccine Communication Strategy

INTERVENTIONS:
Other: HPV Vaccine Communication Strategy — The intervention will include health promotions materials and provision of HPV vaccine

SUMMARY:
Human Papillomavirus (HPV) is the most common sexually transmitted infection globally, and is causally linked to cervical, anogenital, and oropharyngeal cancers. HPV-associated cancers have a disproportionate impact in low-resource settings and nowhere is this evident than in South Africa, which has a uniquely vulnerable population due to the convergence of the largest HIV epidemic globally, with HPV rates of up to 85% in young women under the age of 25. For the clinical trial phase of this study, we intend to evaluate preliminary effects of a communications strategy and key criteria to advance to a full scale hybrid type 2 trial. Our systems-focused approach leverages established partnerships with area schools serving diverse populations who are not always effectively served by traditional healthcare channels.

ELIGIBILITY:
Inclusion Criteria:

* This study will include children enrolled in Grade 5 in participating schools (ages 9-12 years old) in Gauteng province, South Africa, who have no prior history of HPV immunization. We have selected fifth graders for our target population to follow the current Provincial Guidelines. This is in line with National Cervical Guidelines aimed at reaching young people prior to their sexual debut.

We will also be recruiting parents/caregivers of these children, given their role in decision-making. All parents/caregivers will be at least 18 years old. We will also be including adults who are at least 18 years of age, who are employed at participating schools as teachers or school administrators, and others who are engaged in the planning or implementation of the school-based HPV vaccine program (e.g., representatives from the Department of Health, nurses). We have no upper age limit for this population.

Exclusion Criteria:

* Children below the age of 9 years old will not be included in the study.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Uptake of HPV vaccine | within Six Months
  Successful uptake of 1 dose of HPV vaccine
Feasibility of delivering the intervention | Six Months
  Feasibility will be assessed using the Feasibility of Intervention Measure.

SECONDARY OUTCOMES:
Preliminary Effectiveness of the HPV intervention | Six Months
  We will assess HPV vaccine completion at six months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Witwatersrand Health Consortium, Johannesburg, Gautang, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centers for Disease Control and Prevention. Genital HPV Infection - Basic Fact Sheet. 2022. https://www.cdc.gov/std/hpv/stdfact-hpv.htm
- [Background] Szymonowicz KA, Chen J. Biological and clinical aspects of HPV-related cancers. Cancer Biol Med. 2020 Nov 15;17(4):864-878. doi: 10.20892/j.issn.2095-3941.2020.0370. Epub 2020 Dec 15. PMID 33299640
- [Background] South Africa: Human Papillomavirus and Related Cancers, Fact Sheet 2021. Institut Català d'Oncologia; 2021. https://hpvcentre.net/statistics/reports/ZAF_FS.pdf
- See also: South Africa: Human Papillomavirus and Related Cancers, Fact Sheet 2021 by Institut Català d'Oncologia — https://hpvcentre.net/statistics/reports/ZAF_FS.pdf